CLINICAL TRIAL: NCT04660708
Title: Effect of Manual Pelvic Floor Physical Therapy During Pregnancy on Perineal Trauma and Pain in the Post Partum Period
Brief Title: Manual Physical Therapy During Pregnancy on Post Partum Perineal Trauma and Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: Revitalize Physical Therapy (Unknown)
Responsible Party: Principal Investigator, Wendy Huddleston, Associate Professor, University of Wisconsin, Milwaukee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20.102
Record Dates: First submitted 2020-11-04; First posted 2020-12-09 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy Related; Delivery; Injury, Maternal; Pelvic Floor Disorders
Keywords: Manual therapy; physical therapy; post partum
MeSH Terms: conditions — Wounds and Injuries; Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: single-cohort quasi-experimental longitudinal interventions study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women (Experimental): Physical assessment for women 20-34 weeks gestation including evaluating pain, back and hip range of motion, strength of hip and abdominal muscles, diastasis recti, and strength, amount of scar tissue from previous pregnancies / deliveries, level of muscle overactivity, and the extent of any prolapse of pelvic floor muscles.
  Treatment: internal and external myofascial release of the pelvic floor muscles, pelvic floor stretching, and instruction diaphragmatic breathing and exercises for postpartum recovery to perform at home. Exercises include: Pelvic floor stretching: happy baby stretch, deep squat, butterfly stretch; Belly breathing; transverse abdominis contraction, transverse abdominis march, bridge, shoulder blade; Instruction and education on perineal massage and posture.
  Interventions: Behavioral: manual physical therapy

INTERVENTIONS:
Behavioral: manual physical therapy — Previously described in the arm description

SUMMARY:
The purpose of this study is to explore the impact of pelvic floor physical therapy during pregnancy on delivery and the impact on the woman's body and function. Currently there have not been any studies to our knowledge that have examined this relationship and the outcomes for the pregnant patient. The current research that is available is on pelvic floor training and perineal massage during pregnancy with positive outcomes. The questions we are looking to answer include:

1. Does pelvic floor physical therapy during pregnancy decrease the severity of perineal trauma during delivery?
2. Does pelvic floor physical therapy during pregnancy decrease the length of the second stage of labor (pushing)?
3. Does pelvic floor physical therapy during pregnancy decrease the occurrence of emergency C-section?

DETAILED DESCRIPTION:
The purpose of this study is to explore the impact of pelvic floor manual physical therapy techniques during pregnancy on delivery and the impact on the woman's body and function. Currently there have not been any studies to our knowledge that have examined this relationship and the outcomes for the pregnant patient. The current research that is available is on pelvic floor training and perineal massage during pregnancy with positive outcomes. Perineal massage is a stretching technique utilized to relax the tissue of the perineum (the area between the vaginal opening and anus), and is considered routine physical therapy standard of care for pregnant women. Myofascial release of the pelvic floor is a specific manual therapy technique to relax the muscles of the pelvic floor which can include the superficial perineal area. Pelvic myofascial release is a technique used for both pregnant women, and women with chronic pelvic pain. In fact, each component of assessment and treatment are routine and standard PT practices (evaluation, manual therapy, exercise, education), however this specific manual therapy treatment protocol has not been studied during pregnancy to assess the benefits on delivery/recovery. The questions we are looking to answer include:

1. Does pelvic floor PT (physical therapy) during pregnancy decrease the severity of perineal trauma during delivery?
2. Does pelvic floor PT during pregnancy decrease the length of the second stage of labor (pushing)?
3. Does pelvic floor PT during pregnancy decrease the occurrence of emergency C-section?
4. Does pelvic floor PT during pregnancy decrease the likelihood and/or severity of postpartum pelvic pain and pelvic dysfunction? By obtaining these findings, it will allow for program design and treatment recommendations within the pregnancy period to minimize delivery trauma and risk for the mother.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women (any pregnancy, first or subsequent) planning for a vaginal delivery
2. 28-34 weeks gestation at the start of treatment

Exclusion Criteria:

1. Planned c-section
2. < 18 years old
3. >34 weeks gestation
4. Women on pelvic rest

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life and Symptoms Distress Inventory | 7 weeks
  standardized survey to assess level of urinary leakage post partum (0-45 with the higher score indicating greater impairment
Pregnancy Mobility Index | 7 weeks
  standardized survey to determine functional mobility post partum (0 - 72 with a higher score indicating greater impairment)
Delivery type | 7 weeks
  natural or cesarean section (categorical data)
Length of labor | 7 weeks
  length of labor measured in hours
Amount of perineal tearing | 7 weeks
  measured in cm

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Heinecke, DPT, Principal Investigator — Revitalize Physical Therapy
Locations (1):
- Revitalize Physical Therapy, Hales Corners, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No